CLINICAL TRIAL: NCT01711073
Title: Mobilization of Stem Cells With G-CSF and Mozobil in Patients With End Stage Liver Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Proteonomix, Inc. (Industry)
Collaborators: University of Medicine and Dentistry of New Jersey (Other); Numoda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prot001
Record Dates: First submitted 2012-10-11; First posted 2012-10-22 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: End Stage Liver DIsease
MeSH Terms: conditions — End Stage Liver Disease | interventions — Granulocyte Colony-Stimulating Factor; plerixafor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mobilization with G-CSF plus Mozobil (Experimental): Patients will receive G-CSF (Filgrastim) plus Mozobil (Plerixafor)
  Interventions: Drug: Mobilization with G-CSF and Mozobil

INTERVENTIONS:
Drug: Mobilization with G-CSF and Mozobil — Treatment with drugs for mobilization of MSCs
  Other Names: Filgrastim; Neupogen; Plerixafor; AMD3100

SUMMARY:
A phase I trial to study the safety of mobilization of stem cells with G-CSF and Mozobil in patients with chronic liver disease.

DETAILED DESCRIPTION:
Liver cirrhosis in humans represents the end stage of chronic liver injury. Supply of "new" stem cells to the liver could regenerate hepatocytes and restore the lost function. Delivery of Mesenchymal Stem Cells (MSCs) has been shown in animal models and limited clinical trials to result in improved liver disease (MELD) score.

In preclinical studies we have demonstrated that the combination of G-CSF plus Mozobil can effectively mobilize both hematopoietic stem cells (HSCs) and MSCs into the peripheral circulation. While G-CSF only mobilizes HSCs.

The clinical trial will test the safety of treating patients with end stage liver disease with G-CSF and Mozobil to mobilize MSCs into the peripheral circulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of cirrhosis Age greater than or equal to 18 years MELD score less than or equal to 12 able to provide informed consent HIV and HBsAg seronegative Platelet count >50,000, WBC count > 2,000 No history of malignancy within the last 5 years, except for non-melanoma skin cancer or cervical carcinoma in situ No lesions suspicious for liver cancer on CT and/or MRI within prior 4 months

Exclusion Criteria:

Patients with acute or subacute onset of liver disease Patients who have received a liver transplant Age < 18 MELD score >12 Patients whose MELD scores are currently less than or equal to 12 but with history of prior deterioration with MELD score >12 Unable to provide informed consent Patients with HIV or HBsAg seropositivity Pregnant or lactating females Enrolled in another research protocol Any condition that precludes serial follow up Patients with history of malignancy within the last 5 years, except for non-melanoma skin cancer or cervical carcinoma in situ Any lesions suspicious for liver cancer on CT and/or MRI within prior 4 months Patients with palpable splenomegaly on physical examination ANy condition that in the investigators opinion would likely increase the risk of particpation or would likely confound interpretation of the data

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Toxicity as measured by bone pain, hematologic parameters, GI measures and renal parameters | 12 months
  The primary end point for this study is the safety of mobilization of stem cells in patients with end stage liver disease. Adverse events will be documented to assess safety.

SECONDARY OUTCOMES:
Effects of Mobilization | 12 months
  The secondary objective is to study the mobilization of stem cells, including MSCs, to the peripheral circulation and the effect on liver function. Functional assays will define the levels of heamtopoietic stem cells (CD34+ cells) and MSCs (CFU-F) in the circulation of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Baburao Koneru, MD, Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (1):
- University of Medicine and Dentistry of New Jersey, Newark, New Jersey, United States